CLINICAL TRIAL: NCT01847755
Title: Phase 1-2 Study of Hyperbaric Treatment of Traumatic Brain Injury
Brief Title: Hyperbaric Treatment of Traumatic Brain Injury (TBI)
Acronym: TBI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barry Miskin, MD (Other)
Collaborators: Jupiter Medical Center (Other)
Responsible Party: Sponsor-Investigator, Barry Miskin, MD, Principal Investigator, Jupiter Medical Center
Organization: Jupiter Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMC-TBI-001; 117686 (Other: FDA IND application number)
Record Dates: First submitted 2013-04-30; First posted 2013-05-07 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 120 Hyperbaric treatments at 1.5 ATA (Experimental): Patient receives 120 treatments of Hyperbaric at 1.5 ATA. Non randomized trial. Pt will have cognitive assessments and Spect scans at various treatment points. Oxygen is at 1.5 atmospheric pressure.
  Interventions: Drug: Oxygen at 1.5 ATA (atmospheres absolute).

INTERVENTIONS:
Drug: Oxygen at 1.5 ATA (atmospheres absolute). — Each patient will undergo 5 times-a-week Hyperbaric treatments to 1.5 ATA (atmospheres absolute) for up to 120 treatments. Treatment in hyperbaric chamber will be approximately 60 minutes. At specified intervals 40,80,120, patient will be assessed by Spect scan and cognitive assessments to provide outcome measure data. Pt will have a 3 month post treatment follow up assessment.
  Other Names: 02 or Oxygen

SUMMARY:
This study is designed to test the hypothesis that patients with Traumatic Brain Injury (TBI)treated with Hyperbaric (HBO) will show improvement in function and an increased blood flow as evidenced by single-photon emission computerized tomography (SPECT) scan. Improvement is evidenced by increase in number of pixels on SPECT Scan and increased brain metabolism. Improvement may also be identified via cognitive assessments administered by Jupiter Medical Center Research Department.

DETAILED DESCRIPTION:
Patients with Traumatic Brain Injury (TBI)have abnormal findings including hemorrhagic cortical contusions or petechial or foci of altered signal that represents white matter injury. MRI, CT or SPECT scans showing changes consistent with Traumatic Brain Injury (TBI)and or medical history of Traumatic Brain Injury (TBI)as evidenced by medical records will be screened for treatment with Hyperbaric. Each patient will undergo 5 times-a-week Hyperbaric treatments to 1.5 atmospheres absolute(ATA).

Each patient will have a SPECT scan, cognitive assessment, and physician evaluation prior to first treatment and after 40, 80, and 120 treatments to document progress of the treatment (Harch et al, 2012). Cognitive assessment will include the Trail Making Test Parts A and B. Patient will be seen by physician to assess level of disability at each interval; the United States Department of Veteran Affairs' Evaluation of Cognitive Impairment and Subjective Symptoms (VAECI) (2012) tool will be utilized during the physician's evaluation as an objective measure of the patient's level of disability.

Hyperbaric treatments may be adjusted for patient comfort. If the SPECT scan, cognitive assessment and physician evaluation show improvement after 40 treatments, another 40 Hyperbaric(HBO)treatments will be administered. Treatments will be discontinued after a 40 session interval if the SPECT scan, cognitive assessment and physician evaluation show no improvement. The patient will also have a SPECT scan and cognitive assessment follow up 3 months after final Hyperbaric(HBO) treatment.The time points for evaluation of cognitive status and single-photon emission computerized tomography (SPECT) scan will be at at 40,80,120 Hyperbaric(HBO)treatments. Treatment will occur 5 times per week for approximately 24 weeks with another follow up 3 months post treatment. This will provide all data points for outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* All Stage Traumatic Brain Injury (TBI)as demonstrated by loss of consciousness due to the injury that is a minimum of 1 year old
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Women: Negative pregnancy test: If sexually active, women will take contraceptive measures for the duration of the treatments. Medically acceptable contraceptives include: 1) surgical sterilization (such as tubal ligation, hysterectomy, 2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), 3) barrier methods (such as a condom or diaphragm) used with a spermicide, or 4) an intrauterine device (IUD).
* Subjects capacity to give legally effective consent (patient is alert and oriented x3).
* Signed consent form approved by the Institutional Review Board prior to patient entry
* History of lung disease (e.g. bronchitis, asthma) requires chest x-ray prior to inclusion in the study

Exclusion Criteria:

* Untreated Pneumothorax

  * Anti-metabolites/chemotherapeutic agents (is used currently)
  * Mafenide Acetate (sulfamylon): antibacterial drug; peripheral vasodilation Disulfiram (Antabuse)
  * History of spontaneous pneumothorax
  * Seizure Disorder
  * Acute Upper Respiratory Infection
  * Acute High Fever
  * Acute Viral Infection
  * Participation in another experimental trial with active interventions
  * Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Miskin, MD, Principal Investigator — Jupiter Medical Center
Locations (1):
- Jupiter Medical Center, Jupiter, Florida, United States

REFERENCES:
- [Background] Harch PG, Andrews SR, Fogarty EF, Amen D, Pezzullo JC, Lucarini J, Aubrey C, Taylor DV, Staab PK, Van Meter KW. A phase I study of low-pressure hyperbaric oxygen therapy for blast-induced post-concussion syndrome and post-traumatic stress disorder. J Neurotrauma. 2012 Jan 1;29(1):168-85. doi: 10.1089/neu.2011.1895. Epub 2011 Nov 22. PMID 22026588

RESULTS

PARTICIPANT FLOW:
Groups:
- 120 Hyperbaric Treatments at 1.5 ATA: Patient receives 120 treatments of Hyperbaric at 1.5 ATA. Non randomized trial. Pt will have cognitive assessments and Spect scans at various treatment points. Oxygen is at 1.5 atmospheric pressure.
  Oxygen at 1.5 ATA (atmospheres absolute).: Each patient will undergo 5 times-a-week Hyperbaric treatments to 1.5 ATA (atmospheres absolute) for up to 120 treatments. Treatment in hyperbaric chamber will be approximately 60 minutes. At specified intervals 40, 80, 120, patient will be assessed by Spect scan and cognitive assessments to provide outcome measure data. Pt will have a 3 month post treatment follow up assessment.
Period: Overall Study
Arm/Group | 120 Hyperbaric Treatments at 1.5 ATA
Started | 18
Completed | 13
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | 120 Hyperbaric Treatments at 1.5 ATA
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Cerebral Perfusion
Description: This study is designed to test the hypothesis that patients with TBI treated with HBO will show improvement in function and an increased blood flow as evidenced by single-photon emission computerized tomography (SPECT) scan. Improvement is evidenced by increase in number of pixels on SPECT scan and increased brain metabolism.
Time Frame: At 120 Hyperbaric Treatments (5 treatments a week) over approximately 24 weeks with a follow up 3 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 120 Hyperbaric Treatments at 1.5 ATA
Number analyzed (Participants) | 13
Participants | 8

ADVERSE EVENTS:
Time Frame: Approximately 10 months
Arm/Group | 120 Hyperbaric Treatments at 1.5 ATA
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 120 Hyperbaric Treatments at 1.5 ATA (N=18)
Hospitalization (Cardiac disorders) | 1 — Hospitalized due to Hypertension

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT01847755/Prot_SAP_000.pdf